CLINICAL TRIAL: NCT02312544
Title: A Prospective, Multicenter, Randomized, Double-Masked, Parallel-Arm Phase 2b Study Evaluating the Safety and Efficacy of OTX-TP Compared to Timolol Drops in the Treatment of Subjects With Open Angle Glaucoma or Ocular Hypertension
Brief Title: Phase 2b Study Evaluating Safety and Efficacy of OTX-TP Compared to Timolol Drops in the Treatment of Subjects With Open Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ocular Therapeutix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OTX-13-004
Record Dates: First submitted 2014-12-04; First posted 2014-12-09 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-12

CONDITIONS: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Timolol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- OTX-TP treatment (Active Comparator): OTX-TP (sustained release travoprost, 0.36 mg) to be used in this trial with placebo drops administered separately
  Interventions: Drug: OTX-TP
- Timolol control (Active Comparator): Timolol Maleate Ophthalmic Solution, 0.5% dosed twice daily (BID) in the presence of a placebo vehicle punctum plug (PV).
  Interventions: Drug: Timolol

INTERVENTIONS:
Drug: OTX-TP — OTX-TP and placebo drops
  Arms: OTX-TP treatment
Drug: Timolol — Timolol drops and placebo punctum plug
  Arms: Timolol control

SUMMARY:
To evaluate the safety and IOP lowering efficacy of OTX-TP, a sustained release travoprost drug product, placed in the canaliculus of the eyelid compared to Timolol Maleate Ophthalmic Solution, 0.5% in the treatment of subjects with open angle glaucoma or ocular hypertension. The study is designed to assess clinically meaningful response to treatment and is not powered to measure any efficacy endpoints with statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have a documented diagnosis of ocular hypertension, open angle glaucoma (with or without pseudoexfoliation or pigment dispersion component).
* Subject has a mean baseline IOP following washout in at least 1 eye (the same eye) of

  ≥ 24mmHg at Hour 0 (T0) at Baseline Visit 1 and Baseline Visit 2 (Day 1)
* Subject has a mean baseline IOP following washout in at least 1 eye (the same eye) of:

  ≥ 22mmHg at (T0 + 4h) and (T0 + 8h) at Baseline Visit 1 (note: the same eye must meet the IOP eligibility criteria at all 4 baseline assessments)
* Washout IOP must be ≤ 34mmHg in each eye at all time points at the Baseline Visit 1 and Baseline Visit 2 (Day 1)

Exclusion Criteria:

* Subject with any form of glaucoma other than open angle glaucoma (with or without a pigment dispersion or pseudoexfoliation component).
* Subject with mean baseline IOP >34 mmHg in either eye at any time point during the Baseline Visits 1 or 2 (Day 1).
* Subject with a BCVA worse than 0.6 logMAR (20/80 Snellen) in either eye as measured using an ETDRS chart.
* Subject with a known or suspected allergy and/or hypersensitivity to travoprost, timolol, fluorescein or to any component of the study products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2014-11; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Difference in the mean change from baseline average diurnal IOP between treatment groups at the Day 60 Visit | Days 57 to 63
Difference in the mean change from baseline average diurnal IOP between treatment groups at the Day 90 Visit | Days 87 to 93
Difference in the mean change from baseline IOP between treatment groups to each individual time point at the Day 60 and 90 Visits | Days 57 to 63 and Days 87 to 93
Difference in mean IOP between treatment groups for the average diurnal IOP and to each individual time point at the Day 60 and 90 Visits | Days 57 to 63 and Days 87 to 93
Difference in the mean percent change from baseline IOP between treatment groups for the average diurnal IOP and to each individual time point at the Day 60 and 90 Visits | Days 57 to 63 and 87 to 93

CONTACTS AND LOCATIONS:
Locations (1):
- Vold Vision, Fayetteville, Arkansas, United States